CLINICAL TRIAL: NCT00705822
Title: Combination of Docetaxel + Estramustine + Hydrocortisone Versus Docetaxel + Prednisone in Patients With Advanced Prostate Cancer Who Have Relapse in Biochemistry Whilst Androgenic Blockage
Brief Title: Combination of Docetaxel + Estramustine + Hydrocortisone Versus Docetaxel + Prednisone in Patients With Advanced Prostate Cancer
Acronym: PROSTATA
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: low recruitment rate
Sponsor: Sanofi (Industry)
Responsible Party: Medical Affairs Study Director, sanofi-aventis
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: XRP6976J_3502; EudraCT #: 2004-003885-14
Record Dates: First submitted 2008-06-24; First posted 2008-06-26 (Estimated); Last update posted 2010-11-30 (Estimated); Status verified 2010-11

CONDITIONS: Prostatic Neoplasms
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Docetaxel; Estramustine; Hydrocortisone; Prednisone

ARMS (2):
- 1 (Experimental): Docetaxel + Estramustine + Hydrocortisone
  Interventions: Drug: Docetaxel + Estramustine + Hydrocortisone
- 2 (Active Comparator): Docetaxel + Prednisone
  Interventions: Drug: Docetaxel + Prednisone

INTERVENTIONS:
Drug: Docetaxel + Estramustine + Hydrocortisone — Docetaxel iv 80 mg + Oral estramustine-pills 140 mg + Oral hydrocortisone-pills 20 mg.
  Combination of these 3 drugs every 3 weeks
  Arms: 1
Drug: Docetaxel + Prednisone — Docetaxel iv 80 mg + oral prednisone-pills 5 mg. Combination of these 2 drugs every 3 weeks.
  Arms: 2

SUMMARY:
To compare the efficacy of both strategies (reference treatment: Docetaxel+Prednisone and experimental treatment: Docetaxel+Estramustine+Hydrocortisone) by means of PSA values.

To determine the time to treatment failure in both strategies To determine the overall and specific cause survival To evaluate the safety profile To analyze the Quality of Life

ELIGIBILITY:
Inclusion Criteria:

* Histological or cytological confirmation of prostate adenocarcinoma
* Advanced prostate carcinoma.
* Previous treatment with hormones
* Levels of testosterone < 50 ng/dL
* Good hematological, liver and kidney function
* Previous treatment with surgery or radiotherapy, at least 4 weeks since end of treatment is allowed (the patient should have been recovered from any side effects.

Exclusion Criteria:

* Previous chemotherapy (estramustine included).
* Second line hormonotherapy (oestrogens, gestagens, ketoconazole, ...included)
* Previous treatment with radiotherapy (isotopes) or previous radiotherapy over > 25% of the marrow
* Any malignant process with a free disease interval under 5 years, exception done to non-melanoma skin cancer.
* Concomitant serious diseases
* Concomitant treatment with any other neoplassic therapy (exception done to LHRH agonists and/or biphosphonates).
* Contraindication for the treatment with estramustine.
* Previous history of pulmonary embolism, thromboembolic disease, previous treatment with anticoagulants (except aspirin), active thrombophlebitis or hypercoagulation.
* Previous history of pulmonary spillage or ascitis.

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Ages: 18 Years to 75 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2006-08; Primary Completion 2009-07 (Actual); Study Completion 2009-07 (Actual)

PRIMARY OUTCOMES:
Response rate over 50% in PSA | every 3 weeks up to end of treatment and every month until PSA progression

SECONDARY OUTCOMES:
Time to treatment failure | from Informed Consent signature up to end of the study
Time to progression | from Informed Consent signature up to study end
Overall and specific cause surveillance | from Informed Consent signature up to study end
Toxicity profile | from Informed Consent signature up to study end
Patients' Quality of Life | Before first cycle, every 2 cycles throughout the treatment period, at the study end and first follow-up visit

CONTACTS AND LOCATIONS:
Overall Officials: José Taboada, Study Director — Sanofi
Locations (1):
- Sanofi-Aventis Administrative Office, Barcelona, Spain